CLINICAL TRIAL: NCT03739970
Title: A Clinical Trial of Silk Peptide for the Evaluation of Efficacy on Immune Function Enhancement
Brief Title: A Clinical Trial of Silk Peptide for the Evaluation of Efficacy on Immune Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Jong Ho Lee, Professor, Principal Investigator, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 201709-HR-763
Record Dates: First submitted 2018-10-31; First posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Normal Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Group- Silk Peptide (Experimental): * Ingredient: Silk Peptide
  * Type: Yellow granule stick
  * Weight: Silk Peptide 9g/day
  * Directions: with water before breakfast and dinner, 9g/day (4.5g×2times/day)
  * Duration of use: 8 weeks
  Interventions: Dietary Supplement: Investigational Product (Silk Peptide)
- Control Group - Placebo Product (Placebo Comparator): * Ingredient: Microcrystalline Cellulose
  * Type: Yellow granule stick
  * Weight: Silk Peptide 0g/day
  * Directions: with water before breakfast and dinner, 9g/day (4.5g×2times/day)
  * Duration of use: 8 weeks
  Interventions: Dietary Supplement: Control Group - Placebo Product

INTERVENTIONS:
Dietary Supplement: Investigational Product (Silk Peptide) — * Ingredient: Silk Peptide
  * Type: Yellow granule stick
  * Storage: Room temperature
  * Weight: Silk Peptide 9g/day
  * Directions: with water before breakfast and dinner, 9g/day (4.5g×2times/day)
  * Duration of use: 8 weeks
  Arms: Investigational Group- Silk Peptide
Dietary Supplement: Control Group - Placebo Product — * Ingredient: Microcrystalline Cellulose
  * Type: Yellow granule stick
  * Storage: Room temperature
  * Weight: Silk Peptide 0g/day
  * Directions: with water before breakfast and dinner, 9g/day (4.5g×2times/day)
  * Duration of use: 8 weeks
  Arms: Control Group - Placebo Product

SUMMARY:
This study is a 8-week, randomized, double-blind, placebo-controlled clinical trial of Silk Peptide for the evaluation of efficacy on immune function enhancement.

DETAILED DESCRIPTION:
This study will evaluate Silk Peptide's efficacy on immune function in healthy volunteers who white blood cells count is in between 4000/㎕ and 8000/㎕ by assessing improvements in certain immune indices (i.e. NK cell activity, IFN-γ, TNF-α, IL-1β, 2, 12, IgG1, IgG2).

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and female volunteers over 50 years
2. Screening result for WBC counts in between 4,000 cells/ul and 8,000 cells/ul
3. Volunteers who have agreed to participate in the study and provided a written content by him/herself or through its legal representative

Exclusion Criteria:

1. Those with a history of drug and clinically significant hypersensitivity reactions
2. Those with thyroid or pituitary disease
3. Those with acute severe cardiovascular disease such as heart failure, myocardial infarction, and stroke
4. Those with immune system disease or severe liver failure, kidney failure or history
5. Those with a history of systemic diseases such as malignancy, lung disease, leukemia, collagenosis, multiple sclerosis, allergic skin disease and other autoimmune diseases
6. Those with a BMI of less than 18.5 kg/m2 at screening
7. Those diagnosed with diabetes
8. Those with a history of gastrointestinal disorders (ex. Crohn's disease) or gastrointestinal surgery (excluding simple appendectomy or hernia surgery) that may affect the absorption of clinical trial products
9. Those who have consumed medicines, healthy functional foods within 2 weeks before screening or are currently consuming health supplements that can affect immune function. (For health functional foods, they can participate through 1 week before the first intake day.)
10. Those who have received antipsychotic medication within 2 months before screening
11. Those with a alcoholism or history of substance abuse
12. Those who participated in other clinical trials within 2 months before screening
13. Those who are pregnant, breastfeeding
14. Fertile women who do not accept the appropriate method of contraception (except for women who have undergone sterilization operation)
15. Those who are deemed inappropriate by the researcher

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-11-15 (Estimated); Primary Completion 2019-01-29 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
NK(Natural killer) cell activity | 0 week, 8 week
  Changes of NK(Natural killer) cell activity were before and after the intervention

SECONDARY OUTCOMES:
IFN-γ | 0 week, 8 week
  Changes of IFN-γ were before and after the intervention
TNF-α | 0 week, 8 week
  Changes of TNF-α were before and after the intervention
IL-1β | 0 week, 8 week
  Changes of IL-1β were before and after the intervention
IL-2 | 0 week, 8 week
  Changes of IL-2 were before and after the intervention
IL-6 | 0 week, 8 week
  Changes of IL-6 were before and after the intervention
IL-12 | 0 week, 8 week
  Changes of IL-12 were before and after the intervention
IgG1 | 0 week, 8 week
  Changes of IgG1 were before and after the intervention
IgG2 | 0 week, 8 week
  Changes of IgG2 were before and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: JONGHO LEE, Ph.D., Principal Investigator — Yonsei University
Locations (1):
- Laboratory of Clinical Nutrigenetics/Nutrigenomics, Yonsei University., Seoul, South Korea